CLINICAL TRIAL: NCT04022564
Title: Incidence, and Survival Medical Expenditure of Patients With Multiple Sclerosis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Chun-Ming Liao (Other)
Responsible Party: Sponsor-Investigator, Chun-Ming Liao, Project Manager, China Medical University Hospital
Organization: China Medical University Hospital (Other)
Other Study IDs: CMUH108-REC2-084
Record Dates: First submitted 2019-07-15; First posted 2019-07-17 (Actual); Last update posted 2019-07-17 (Actual); Status verified 2019-07

CONDITIONS: Neurologic Signs and Symptoms
Keywords: multiple sclerosis; Survival Analysis; cause of death; medical resources
MeSH Terms: conditions — Neurologic Manifestations; Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- The subjects are diagnosed as MS patient: The study population is based on the 'National Health Insurance Research Database' (NHIRD) from 2001 to 2015 provided by Taiwan Ministry of Health and Welfare. The subjects are diagnosed as MS patients based on the 'Registry for Catastrophic Illness'.

SUMMARY:
Multiple sclerosis (MS) is a disease of autoimmune system which attacks the central nervous system and that is one of the most common inflammatory diseases and has caused a heavy disease burden on patients. In the world, the prevalence of MS is on the rise, and the annual growth rate of MS patients in Taiwan is much higher than the whole world (3.78 times). However, it has no discussion or study in references at present, and it is worthwhile to research. MS is not a fatal disease, but its complications make the mortality of its patients three times higher than that of general population. This study will explore the survival and the causes of death for MS patients in Taiwan by cohort study of fourteen years. In addition, in the recent years, the MS patients in Taiwan and the medical resource consumption has increased largely, and it is necessary to conduct the research.

DETAILED DESCRIPTION:
The study population is based on the 'National Health Insurance Research Database' (NHIRD) from 2001 to 2015 provided by Taiwan Ministry of Health and Welfare. The subjects are diagnosed as MS patients based on the 'Registry for Catastrophic Illness'. First, the investigators will perform the statistical analysis of the incidence, the prevalence, the mortality and the trend analysis of the MS patients diagnosed each year. First, Kaplan-Meier method will be employed to examine the survival curves. Next, Cox proportional hazards model will be used to analyze the survival and related factors. Last, multiple regression analysis will be then performed to analyze the influence of independent variables on patients' medical utilization in each year.

In response to the lack of data on population-based epidemiological studies on MS diseases in Asia, this research wishes to fill the gaps in the studies of global prevention and analyze the patient's survival, mortality risk factors and the medical utilization as a reference for national health policies.

ELIGIBILITY:
Inclusion Criteria:

* The subjects are diagnosed as MS patients

Exclusion Criteria:

* The subjects are not diagnosed as MS patients

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population is based on the 'National Health Insurance Research Database' (NHIRD) from 2001 to 2015 provided by Taiwan Ministry of Health and Welfare.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2019-07-15 (Actual); Primary Completion 2020-05-20 (Estimated); Study Completion 2020-05-20 (Estimated)

PRIMARY OUTCOMES:
Incidence, and SurvivalMedical Expenditure of Patients with Multiple Sclerosis | 'National Health Insurance Research Database' (NHIRD) from 2001 to 2015
  we will perform the statistical analysis of the incidence, the prevalence, the mortality and the trend analysis of the MS patients diagnosed each year. First, Kaplan-Meier method will be employed to examine the survival curves. Next, Cox proportional hazards model will be used to analyze the survival and related factors. Last, multiple regression analysis will be then performed to analyze the influence of independent variables on patients' medical utilization in each year.

CONTACTS AND LOCATIONS:
Locations (1):
- Genetic and Rare Disease Center, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No